CLINICAL TRIAL: NCT03276117
Title: Wide Using of Paperless Partograph in Evaluation of Labour
Brief Title: Wide Use of Paperless Partograph in Evaluation of Labour
Acronym: labourRecord
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, ayman darder, principal investigator, Assiut University
Other Study IDs: paperless partograph
Record Dates: First submitted 2017-09-04; First posted 2017-09-08 (Actual); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: Labor Complication; Labor Pain
Keywords: pregnancy.obstructed labour
MeSH Terms: conditions — Obstetric Labor Complications; Labor Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Inside labour room we record that when the labour women in active phase as cervical dilatation 4cm or more
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Paperless partograph wide using in labour room as simple tool in evaluation of labour

DETAILED DESCRIPTION:
Both world health organization ( WHO) PARTOGRAPH and modified world heath organization (WHO)PARTOGRAPH are too long labour tools in evaluation of labour so we need simple tool in evaluation of labour

ELIGIBILITY:
Inclusion Criteria:

* Spontaneous labour
* cephalic presentation
* pregnant 37 weeks up to full term

Exclusion Criteria:

* mail_presentation
* induced labour

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: the collected data wail be analyzed using the statistical package for social science (version 10.0 for windows,SPSS.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2017-08-21 (Actual); Study Completion 2017-08-26 (Actual)

PRIMARY OUTCOMES:
Progress of labour | up to 2 month
  Cervical dilated 1 cm each hour

SECONDARY OUTCOMES:
New born | up to 1 month
  Apgar scor at 1 minute and Apgar scor at 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: mohamed khalaph, professor, Study Chair — assiut universty faculity of medicine; ahmad abass, professor, Principal Investigator — assiut university faclity of meficibe
Locations (6):
- Egypt (6):
  - Faculity of Medicine ,in Assiut,Egypt, Asyut
  - Faculity of Medicine Assiut University, Asyut
  - Faculity of Medicine in Assiut,Egypt, Asyut
  - Faculity of Medicine,in Assiut ,Egypt, Asyut
  - Faculity of Medicine,in Assiut,Egypt, Asyut
  - Faculity of Medicine, Asyut

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Jadad AR, McQuay HJ. Searching the literature. Be systematic in your searching. BMJ. 1993 Jul 3;307(6895):66. doi: 10.1136/bmj.307.6895.66-a. No abstract available. PMID 8343701
- [Result] Chang AA, Heskett KM, Davidson TM. Searching the literature using medical subject headings versus text word with PubMed. Laryngoscope. 2006 Feb;116(2):336-40. doi: 10.1097/01.mlg.0000195371.72887.a2. PMID 16467730
- [Result] Fatehi F, Gray LC, Wootton R. How to improve your PubMed/MEDLINE searches: 3. advanced searching, MeSH and My NCBI. J Telemed Telecare. 2014 Mar;20(2):102-12. doi: 10.1177/1357633X13519036. PMID 24614997
- See also: all the journals articles are available online to the readers all over the world without legal barriers — http://www.iiste.org/journals/